CLINICAL TRIAL: NCT05590156
Title: Can Action Observation Therapy be an Alternative to Robotic Rehabilitation to Improve Upper Extremity Functions in Stroke Patients? A Protocol of Randomized Controlled Study
Brief Title: Effects of the Action Observation Therapy and Robotic Rehabilitation on the Upper-Limb Motor Function in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Şenocak (Other)
Responsible Party: Sponsor-Investigator, Emre Şenocak, Research Assistant, Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2022.649
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: Robotic Rehabilitation; Action Observation Therapy; Upper Extremity; Motor Function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation Therapy (AOT) (Experimental): AOT is a method based on the principle that the patient watches the movements of a healthy individual and then tries to imitate them. AOT consists of a monitoring-imitation cycle. A cycle consists of 3 minutes of observation, and 3 minutes of imitation. The intervention will consist of 10 cycles for simple functions. Complex movements will be applied by separating them into their components. The cycle time for each component is the same. Take for example, the cup-reaching function: The first component is the cup-reaching activity. The second component is the glass grip. One cycle will be completed on the first component (6 minutes), then one cycle will be completed for the second component (6 minutes) and one cycle (6 minutes) will be completed for the entire movement. Cycles will follow each other for 60 minutes.
  For the AOT, 31 different videos were prepared for the shoulder, elbow, and wrist. Applications will be made in the hospital under the supervision of a physiotherapist.
  Interventions: Procedure: Conventional Rehabilitation; Procedure: Action Observation Therapy (AOT)
- Robotic Rehabilitation (Experimental): The robotic rehabilitation application will be performed with the ExoRehab X (HoustonBionics, Inc.) device. There is no engine to create any repulsive-pulling force in this device. It is a system that works entirely with the patient's active movement.
  Active movements of the shoulder, elbow, and wrist in all directions can be performed with the device. Motion is detected with the help of the device's censor, and the avatar moves on the screen. There are 10 different purposeful games embedded in the device. The device also allows resistance exercise thanks to resistance modules.
  Which joint will be trained will be determined according to the potential of the patient. For example, if programming will be done for the shoulder, elbow and wrist, the treatment time will be 20 minutes for each joint.
  Applications will be made in the hospital under the supervision of a physiotherapist.
  Interventions: Procedure: Conventional Rehabilitation; Device: Robotic Rehabilitation (ExoRehab X)

INTERVENTIONS:
Procedure: Conventional Rehabilitation — Conventional treatment for the upper extremity will be applied according to the patient's individual needs. A physiotherapist will apply this method in the clinic for 60 minutes. The duration of treatment is 60x3x8 minutes/day/week. Other methods will be applied in addition to the conventional treatment program.
Device: Robotic Rehabilitation (ExoRehab X) — Robotic Rehabilitation
  Arms: Robotic Rehabilitation
Procedure: Action Observation Therapy (AOT) — Action Observation Therapy (AOT)
  Arms: Action Observation Therapy (AOT)

SUMMARY:
This protocol will investigate the effects of action observation therapy and robotic rehabilitation on upper extremity motor functions in subacute stroke patients. Firstly, for this purpose, conventional rehabilitation approaches will take 60 minutes before both treatment methods in stroke patients. The upper-limb conventional rehabilitation program will be applied to all patients according to their individual needs (60x3x8 minutes/day/week). This program will consist of purposeful clinical exercises with a physiotherapist.

After the conventional rehabilitation, one of the groups will receive action observation therapy, while the other will receive robotic rehabilitation. Both additional treatment methods will also be applied for 60 minutes. Treatment durations of both additional treatments are the same (60x3x8 minutes/day/week). Assessments will be made three times (Beginning, 4th week, 8th week).

DETAILED DESCRIPTION:
Randomization: The online randomization software (www.randomizer.org) will be used for the study. After randomization, patients will be divided into two groups (AOT group, Robotic group)

Blinding: Due to the nature of the study, patient-practitioner blinding is not possible. But an independent expert will perform the statistical analysis, and single-blind will be provided.

Estimating Sample Size: Gpower 3.1.9.7 software was used for sample size calculation. To calculate the effect size, the study of Lima and Christofoletti was taken as a reference, and the effect size was calculated as 1.29. The alpha error was accepted as 5% and the power of the study was 80%. Accordingly, considering that there may be missing data in the study, it was planned to include a minimum of 30 stroke patients.

Statistical Analysis: Statistical Package for the Social Sciences (SPSS v11.5) program will be used for analysis. Whether the data is normally distributed or not will be questioned by the Shapiro-Wilks test and histogram curves. When the data are normally distributed, Independent Sample T-test will be used for comparisons between groups, and Paired-Sample T-test will be used for comparisons within groups. When the data do not show normal distribution, Mann-Whitney U Test will be used for intergroup comparisons and Wilcoxon Signed Rank Test will be used for in-group comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-80 aged
* Stroke history in last six months
* Mini-Mental Status Evaluation >24 points,
* Having an Ability to sit independently,
* Presence of at least half of the range of motion of all joints for the upper extremity,
* Spasticity ≤ 2 according to the Modified Ashworth Scale,
* The Fugl-Meyer Assessment for Upper Extremity score between 20-60,
* Individuals without visual impairment,
* Individuals with normal communication and cooperation skills.

Exclusion Criteria:

* Having another neurological disease,
* Having any orthopedic problems that may affect the upper extremity,
* Taking neuropsychiatric treatment,
* Individuals who had a botox history or tendon surgery,
* Using neuroleptic drugs,
* Having an ataxia,
* Individuals who attended less than 80% of the total number of sessions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment for Upper Extremity | Baseline
  This form is used to detect healing in the upper extremity.
Fugl Meyer Assessment for Upper Extremity | End of the 4th week
  This form is used to detect healing in the upper extremity.
Fugl Meyer Assessment for Upper Extremity | End of the 8th week
  This form is used to detect healing in the upper extremity.
Wolf Motor Function Test | Baseline
  This test is used for the level of motor function.
Wolf Motor Function Test | End of the 4th week
  This test is used for the level of motor function.
Wolf Motor Function Test | End of the 8th week
  This test is used for the level of motor function.

SECONDARY OUTCOMES:
Demographic Data Form | Baseline
  Informations about the patients
Functional Independence questionnaire | Baseline
  This form helps determine an individual's level of independence.
Functional Independence questionnaire | End of the 4th week
  This form helps determine an individual's level of independence.
Functional Independence questionnaire | End of the 8th week
  This form helps determine an individual's level of independence.
The Stroke-Specific Quality of Life Scale (SS-QoL) | Baseline
  This is a quality of life assessment scale specific to stroke patients. Individuals with a high quality of life also have a high score.
The Stroke-Specific Quality of Life Scale (SS-QoL) | End of the 4th week
  This is a quality of life assessment scale specific to stroke patients. Individuals with a high quality of life also have a high score.
The Stroke-Specific Quality of Life Scale (SS-QoL) | End of the 8th week
  This is a quality of life assessment scale specific to stroke patients. Individuals with a high quality of life also have a high score.
Box and Block Test | Baseline
  This test is used to evaluate gross motor function of the upper extremity.
Box and Block Test | End of the 4th week
  This test is used to evaluate gross motor function of the upper extremity.
Box and Block Test | End of the 8th week
  This test is used to evaluate gross motor function of the upper extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Şenocak, MSc, Study Director — Marmara University; Aysel Yildiz Ozer, PhD, Study Chair — Marmara University; Elif Korkut, PhD, Study Director — Bağcılar Education and Research Hospital; Adem Aktürk, PhD, Study Director — İstanbul Gelişim University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No